CLINICAL TRIAL: NCT00382070
Title: A Clinical Trial to Determine the Efficacy of Five Years of Letrozole Compared to Placebo in Patients Completing Five Years of Hormonal Therapy Consisting of an Aromatase Inhibitor (AI) or Tamoxifen Followed by an AI in Prolonging Disease-Free Survival in Postmenopausal Women With Hormone Receptor Positive Breast Cancer
Brief Title: Letrozole in Treating Postmenopausal Women Who Have Received Hormone Therapy for Hormone Receptor-Positive Breast Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NSABP B-42; U10CA012027 (NIH)
Record Dates: First submitted 2006-09-26; First posted 2006-09-28 (Estimated); Results first posted 2021-05-20 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 2 Letrozole (Experimental): Patients receive oral letrozole once daily for up to 5 years.
  Interventions: Drug: Letrozole
- Group 1 Placebo (Placebo Comparator): Patients receive oral placebo once daily for up to 5 years.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Letrozole — Letrozole 2.5 mg taken orally once daily for 5 years
  Arms: Group 2 Letrozole
Other: Placebo — Placebo tablet taken orally once daily for 5 years
  Arms: Group 1 Placebo

SUMMARY:
RATIONALE: Estrogen can cause the growth of breast cancer cells. Hormone therapy using letrozole may fight breast cancer by lowering the amount of estrogen the body makes. It is not yet known whether letrozole is more effective than a placebo in treating patients with hormone receptor-positive breast cancer.

PURPOSE: This randomized phase III trial is studying letrozole to see how well it works compared with a placebo in treating postmenopausal women who have received hormone therapy for hormone receptor-positive breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether or not prolonged adjuvant hormonal therapy comprising letrozole vs placebo will improve disease-free survival of postmenopausal women with estrogen receptor-positive and/or progesterone receptor-positive breast cancer who have completed 5 years of hormonal therapy with 5 years of an aromatase inhibitor (AI) or 5 years of a combination of up to 3 years of tamoxifen citrate followed by an AI.
* Compare the disease-free survival of patients treated with these regimens.

Secondary

* Compare overall survival of patients treated with these regimens.
* Compare breast cancer-free interval of patients treated with these regimens.
* Compare distant recurrence in patients treated with these regimens.
* Compare the incidence of osteoporotic-related fractures (e.g., Colles', hip, and spine) in these patients treated with these regimens.
* Compare the incidence of arterial thrombotic events in patients treated with these regimens.

OUTLINE: This is a double-blind, multicenter, placebo-controlled, randomized study. Patients are stratified according to pathologic nodal status (negative vs positive), adjuvant tamoxifen citrate therapy (yes vs no), and lowest bone mineral density T score for lumbosacral spine, total hip, or femoral neck (> -2.0 vs ≤ -2.0 standard deviation). Patients are randomized to 1 of 2 treatment arms.

* Group I: Patients receive oral placebo once daily.
* Group II: Patients receive oral letrozole once daily.

In both arms, treatment continues for up to 5 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed annually.

PROJECTED ACCRUAL: A total of 3,840 patients will be accrued for this study.

ELIGIBILITY:
Eligibility Criteria

* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (0 = fully active, able to carry on all pre-disease performance without restriction; 1 = restricted in physically strenuous activity but ambulatory).
* Patients must be postmenopausal at the time of randomization. (Note: Premenopausal or perimenopausal women requiring therapy with luteinizing hormone-releasing hormone [LHRH] analogs to suppress ovarian function are not eligible.) For study purposes, postmenopausal is defined as: age 56 or older with no spontaneous menses for at least 12 months prior to study entry, or age 55 or younger with no spontaneous menses for at least 12 months prior to study entry (e.g., spontaneous or secondary to hysterectomy) AND with a documented estradiol level in the postmenopausal range according to local institutional/laboratory standards, or a prior documented bilateral oophorectomy.
* The patient must have remained disease-free from the time of initial breast cancer diagnosis until the time of randomization.
* The patient must have had histologically-confirmed invasive carcinoma of the breast by diagnostic core needle biopsy or by final pathologic evaluation of the surgical specimen.
* Patients who received neoadjuvant chemotherapy must have been clinical Stage I, II, or IIIA. For patients who received adjuvant chemotherapy, the primary tumor must have been T1-3 on pathologic evaluation and ipsilateral nodes must have been pN0, pN1 (pN1mi, pN1a, pN1b, pN1c), pN2a, pN3a, or pN3b.
* The primary tumor must have been estrogen receptor (ER)-positive and/or progesterone receptor (PgR)-positive. (Patients who had a tumor that was considered to be borderline for hormone receptor positivity and who were treated with tamoxifen and/or an aromatases inhibitor (AI) are eligible for this study.)
* Patients must have undergone either a lumpectomy with axillary nodal staging followed by breast radiotherapy or a total mastectomy with axillary nodal staging. (Acceptable axillary nodal staging procedures include sentinel node biopsy alone, if sentinel nodes were negative on hematoxylin and eosin (H&E) staining.)
* The duration of the patient's hormonal therapy following breast cancer diagnosis must have been 57-63 months from the first dose regardless of the number of missed doses. Hormonal therapy must have consisted of an AI or a combination of up to 3 years of tamoxifen followed by an AI. Tamoxifen may not have been given during years 4 and 5 of the 5 years of adjuvant hormonal therapy. (Note: Patients must discontinue their adjuvant AI therapy at the time of randomization.)
* Optional Letrozole Registration Program for patients who have not yet completed 5 years of hormonal therapy. (Note: As of September 5, 2008, the optional NSABP B-42 Registration Program closed to patient enrollment. Accrual and data collection for the NSABP B-42 randomized treatment trial continues as planned.) In order to have a predominantly letrozole-treated population for B-42 study entry, patients who have had a minimum of 2 years of hormonal therapy and who are currently on tamoxifen (for up to 3 years) or an AI may be offered letrozole at no cost until they complete 5 total years of initial adjuvant hormonal therapy.
* B-42 randomization must be within 6 months following completion of 5 years (57-63 months) of initial adjuvant hormonal therapy.
* At the time of randomization, the patient must have had the following: history and physical exam within 3 months demonstrating no findings suggestive of recurrent breast cancer; bilateral mammogram within 1 year (unilateral if patient had a mastectomy); mammogram not required if patient had a prophylactic contralateral mastectomy; bone mineral density (BMD) testing within 1 year; and fasting lipid profile (total cholesterol, LDL-C, HDL-C, and triglycerides) with a total cholesterol value less than or equal to grade 1 (according to CTCAE v3.0), with or without cholesterol-lowering therapy.

  * within 1 year if the patient has a history of hypercholesterolemia controlled with cholesterol-lowering therapy and/or therapeutic lifestyle changes or if the patient has a history of one or more of the following risk factors for future cardiovascular events: diabetes, hypertension, obesity, tobacco use, hypertriglyceridemia, documented coronary artery disease, or family history of premature coronary heart disease.
  * within 2 years for all other patients.

Ineligibility Criteria

* Patients with one or more of the following conditions will be ineligible for this study:
* History of non-traumatic osteoporotic fracture of wrist, hip, or spine.
* Diagnosis of bilateral breast cancer including ductal carcinoma in situ (DCIS)[(synchronous or metachronous].
* Other malignancies unless the patient is considered to be disease-free for 5 or more years prior to randomization, and is deemed by their physician to be at low risk for recurrence. Patients with the following cancers are eligible if diagnosed and treated within the past 5 years: carcinoma in situ of the cervix, colon carcinoma in situ, melanoma in situ, and basal cell and squamous cell carcinoma of the skin.
* Sex hormonal therapy, e.g., estrogen- or progesterone-replacement therapy or oral contraceptives. These patients are eligible only if this therapy is discontinued prior to randomization.
* Therapy with any hormonal agent such as raloxifene for management of osteoporosis. Patients are eligible only if these medications are discontinued prior to study entry.
* Administration of any investigational agent within 30 days before study entry.

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3966 (Actual)
Dates: Start 2006-08; Primary Completion 2016-08-25 (Actual); Study Completion 2025-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (806):
- United States (777):
  - Regional Medical Center, Anniston, Alabama
  - Providence Cancer Center at Providence Hospital, Mobile, Alabama
  - Providence Cancer Center, Anchorage, Alaska
  - Fairbanks Cancer Treatment Center at Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Peninsula Medical Center, Burlingame, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants - Castro Valley, Castro Valley, California
  - Cancer Care Center at John Muir Health - Concord Campus, Concord, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - North Bay Cancer Center, Fairfield, California
  - Kaiser Permanente - Fremont, Fremont, California
  - Valley Medical Oncology, Fremont, California
  - Cancer Care Associates, Fresno, California
  - Virginia K. Crosson Cancer Center at St. Jude Medical Center, Fullerton, California
  - Glendale Memorial Hospital Comprehensive Cancer Center, Glendale, California
  - Marin Cancer Institute at Marin General Hospital, Greenbrae, California
  - Sutter Health - Western Division Cancer Research Group, Greenbrae, California
  - Kaiser Permanente Medical Center - Hayward, Hayward, California
  - Scripps Cancer Center - San Diego, La Jolla, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Breastlink Medical Group, Incorporated at Long Beach Memorial Medical Center, Long Beach, California
  - Pacific Shores Medical Group - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - El Camino Hospital Cancer Center, Mountain View, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Breast Surgeons, Incorporated, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee, Incorporated, Oakland, California
  - Kaiser Permanente Medical Center - Oakland, Oakland, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - St. Joseph Hospital Regional Cancer Center - Orange, Orange, California
  - Desert Regional Medical Center Comprehensive Cancer Center, Palm Springs, California
  - Valley Care Medical Center, Pleasanton, California
  - Valley Medical Oncology Consultants - Pleasanton, Pleasanton, California
  - Robert and Beverly Lewis Family Cancer Care Center at Pomona Valley Hospital Medical Center, Pomona, California
  - Lucy Curci Cancer Center at Eisenhower Memorial Hospital and Medical Center, Rancho Mirage, California
  - North Valley Breast Clinic, Redding, California
  - Kaiser Permanente Medical Center - Redwood City, Redwood City, California
  - Kaiser Permanente Medical Center - Richmond, Richmond, California
  - Kaiser Permanente Medical Center - Roseville, Roseville, California
  - Sutter Cancer Center at Roseville Medical Center, Roseville, California
  - Sutter Cancer Center, Sacramento, California
  - South Sacramento Kaiser-Permanente Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Salinas Valley Memorial Hospital, Salinas, California
  - Kaiser Permanente Medical Office -Vandever Medical Office, San Diego, California
  - San Francisco General Hospital Medical Center, San Francisco, California
  - Kaiser Permanente Medical Center - San Francisco Geary Campus, San Francisco, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Teresa, San Jose, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - Kaiser Foundation Hospital - San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - Kaiser Permanente Medical Center - Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Medical Center - South San Francisco, South San Francisco, California
  - Stanford Cancer Center, Stanford, California
  - Kaiser Permanente Medical Facility - Stockton, Stockton, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Sutter Solano Medical Center, Vallejo, California
  - Kaiser Permanente Medical Center - Walnut Creek, Walnut Creek, California
  - John Muir/Mt. Diablo Comprehensive Cancer Center, Walnut Creek, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Memorial Hospital Cancer Center - Colorado Springs, Colorado Springs, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Shaw Regional Cancer Center, Edwards, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Bristol Hospital, Bristol, Connecticut
  - Praxair Cancer Center at Danbury Hospital, Danbury, Connecticut
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Farmington, Connecticut
  - Helen and Harry Gray Cancer Center at Hartford Hospital, Hartford, Connecticut
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Middlesex Hospital Cancer Center, Middletown, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Carl and Dorothy Bennett Cancer Center at Stamford Hospital, Stamford, Connecticut
  - Connecticut Oncology & Hematology - Torrington, Torrington, Connecticut
  - Harold Leever Regional Cancer Center, Waterbury, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Washington Cancer Institute at Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Eugene M. and Christine E. Lynn Cancer Institute at Boca Raton Community Hospital - West, Boca Raton, Florida
  - Eugene M. and Christine E. Lynn Cancer Institute at Boca Raton Community Hospital - Main Campus, Boca Raton, Florida
  - Morton Plant Hospital, Clearwater, Florida
  - Herbert D. Kerman Regional Oncology Center - Daytona Beach, Daytona Beach, Florida
  - North Broward Medical Center, Deerfield Beach, Florida
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Center for Cancer Care and Research at Watson Clinic, LLP, Lakeland, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Integrated Community Oncology Network - Orange Park, Orange Park, Florida
  - M.D. Anderson Cancer Center at Orlando, Orlando, Florida
  - Florida Cancer Specialists - Sarasota Downtown, Sarasota, Florida
  - Cleveland Clinic Florida - Weston, Weston, Florida
  - Phoebe Cancer Center at Phoebe Putney Memorial Hospital, Albany, Georgia
  - Northeast Georgia Cancer Care, LLC - Medical Oncology, Athens, Georgia
  - Georgia Cancer Center for Excellence at Grady Memorial Hospital, Atlanta, Georgia
  - Emory Crawford Long Hospital, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Augusta Oncology Associates - Walton Way, Augusta, Georgia
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - John B. Amos Cancer Center, Columbus, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Harbin Clinic Cancer Center - Medical Oncology, Rome, Georgia
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - Hawaii Medical Center - East, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute - Maui, Wailuku, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - Kootenai Cancer Center - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Resurrection Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Creticos Cancer Center at Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Sherman Hospital, Elgin, Illinois
  - Alexian Brothers Radiation Oncology, Elk Grove Village, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Evanston Hospital, Evanston, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Provena St. Mary's Regional Cancer Center - Kankakee, Kankakee, Illinois
  - La Grange Memorial Hospital, La Grange, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Edward Hospital Cancer Center, Naperville, Illinois
  - Hematology Oncology Consultants - Naperville, Naperville, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Advocate Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Center for Cancer Care at OSF Saint Anthony Medical Center, Rockford, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Central Dupage Cancer Center, Winfield, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Center for Cancer Care at Goshen General Hospital, Goshen, Indiana
  - Community Regional Cancer Care at Community Hospital East, Indianapolis, Indiana
  - Community Regional Cancer Care at Community Hospital North, Indianapolis, Indiana
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Horizon Oncology Center, Lafayette, Indiana
  - Community Hospital, Munster, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Bettendorf, Iowa
  - Iowa Blood and Cancer Care, Cedar Rapids, Iowa
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Heartland Oncology and Hematology, Council Bluffs, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Genesis Medical Center - West Campus, Davenport, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cedar Valley Medical Specialists, PC - West Ridgeway Avenue, Waterloo, Iowa
  - Covenant Cancer Treatment Center, Waterloo, Iowa
  - Hospital District Sixth of Harper County, Anthony, Kansas
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Mount Carmel Regional Cancer Center, Pittsburg, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Cancer Resource Center at King's Daughters Medical Center, Ashland, Kentucky
  - Cancer Care at Our Lady of Bellefonte Hospital, Ashland, Kentucky
  - Central Baptist Hospital, Lexington, Kentucky
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Louisville Oncology at Norton Cancer Institute - Louisville, Louisville, Kentucky
  - Consultants in Blood Disorders and Cancer, Louisville, Kentucky
  - Drs. Carrol, Sheth, Raghavan, Louisville, Kentucky
  - Pennington Cancer Center at Baton Rouge General, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - Ochsner Health Center - Bluebonnet, Baton Rouge, Louisiana
  - Terrebonne General Medical Center, Houma, Louisiana
  - Drs Gurtler Brinz and Russo APMC-Metairie Oncologists, Metairie, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - Christus Schumpert Cancer Treatment Center, Shreveport, Louisiana
  - CancerCare of Maine at Eastern Maine Medical Center, Bangor, Maine
  - Central Maine Comprehensive Cancer Center at Central Maine Medical Center, Lewiston, Maine
  - Mercy Hospital, Portland, Maine
  - York Hospital's Oncology Treatment Center, York Village, Maine
  - Mercy Medical Center, Baltimore, Maryland
  - Greater Baltimore Medical Center Cancer Center, Baltimore, Maryland
  - St. Agnes Hospital Cancer Center, Baltimore, Maryland
  - Harry & Jeanette Weinberg Cancer Institute at Franklin Square Hospital Center, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - Shore Regional Cancer Center at Memorial Hospital - Easton, Easton, Maryland
  - Union Hospital Cancer Program at Union Hospital, Elkton, Maryland
  - Frederick Memorial Hospital Regional Cancer Therapy Center, Frederick, Maryland
  - St. Mary's Hospital, Leonardtown, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Sturdy Memorial Hospital, Attleboro, Massachusetts
  - Tufts-NEMC Cancer Center, Boston, Massachusetts
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Lahey Clinic Medical Center - Burlington, Burlington, Massachusetts
  - Commonwealth Hematology-Oncology, PC - Concord, Concord, Massachusetts
  - Commonwealth Hematology Oncology PC - Dorchester, Dorchester, Massachusetts
  - Hudner Oncology Center at Saint Anne's Hospital - Fall River, Fall River, Massachusetts
  - Simonds-Sinon Regional Cancer Center at HealthAlliance Hospital - Burbank Campus, Fitchburg, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Commonwealth Hematology-Oncology, PC - Lawrence, Lawrence, Massachusetts
  - Commonwealth Hematology Oncology PC - Leominster, Leominster, Massachusetts
  - Caritas Holy Family Hospital, Methuen, Massachusetts
  - NSMC Cancer Center - Peabody, Peabody, Massachusetts
  - Berkshire Hematology Oncology, PC, Pittsfield, Massachusetts
  - Jordan Hospital Club Cancer Center, Plymouth, Massachusetts
  - Commonwealth Hematology-Oncology, PC - Quincy, Quincy, Massachusetts
  - Baystate Regional Cancer Program at D'Amour Center for Cancer Care, Springfield, Massachusetts
  - Commonwealth Hematology-Oncology, PC - Stoneham, Stoneham, Massachusetts
  - Commonwealth Hematology-Oncology, PC - Weymouth, Weymouth, Massachusetts
  - Commonwealth Hematology-Oncology, PC - Worcester, Worcester, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Bay Regional Medical Center, Bay City, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Great Lakes Cancer Institute at McLaren Regional Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Lapeer Regional Hospital, Lapeer, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Upper Michigan Cancer Center at Marquette General Hospital, Marquette, Michigan
  - MidMichigan Medical Center - Midland, Midland, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Clemens Regional Medical Center, Mount Clemens, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - St. Luke's Hospital Cancer Care Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Immanuel St. Joseph's, Mankato, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Hattiesburg Clinic, PA at Forrest General, Hattiesburg, Mississippi
  - Keesler Air Force Base Medical Center, Keesler Air Force Base, Mississippi
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Freeman Cancer Institute at Freeman Health System, Joplin, Missouri
  - St. John's Regional Medical Center, Joplin, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Midwest Hematology Oncology Group, Incorporated, St Louis, Missouri
  - Saint Louis University Cancer Center, St Louis, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - St. Anthony's Cancer Center, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Arch Medical Services, Incorporated at Center for Cancer Care and Research, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Saint Francis Cancer Treatment Center at Saint Francis Memorial Health Center, Grand Island, Nebraska
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - Callahan Cancer Center at Great Plains Regional Medical Center, North Platte, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - New Hampshire Oncology - Hematology, PA at Payson Center for Cancer Care, Concord, New Hampshire
  - Seacoast Cancer Center at Wentworth - Douglass Hospital, Dover, New Hampshire
  - Center for Cancer Care at Exeter Hospital, Exeter, New Hampshire
  - New Hampshire Oncology - Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Lakes Region General Hospital, Laconia, New Hampshire
  - Portsmouth Regional Hospital, Portsmouth, New Hampshire
  - Ocean Medical Center at Meridian Health, Brick, New Jersey
  - Dizzy Gillespie Cancer Institute at Englewood Hospital and Medical Center, Englewood, New Jersey
  - Hunterdon Regional Cancer Center at Hunterdon Medical Center, Flemington, New Jersey
  - CentraState Medical Center, Freehold, New Jersey
  - Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - St. Barnabas Medical Center Cancer Center, Livingston, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - AtlantiCare Cancer Care Institute at AtlantiCare Regional Medical Center - Mainland Campus, Pomona, New Jersey
  - University Medical Center at Princeton, Princeton, New Jersey
  - Booker Cancer Center at Riverview Medical Center, Red Bank, New Jersey
  - Valley Hospital - Ridgewood, Ridgewood, New Jersey
  - Somerset Medical Center, Somerville, New Jersey
  - Frederick R. and Betty M. Smith Cancer Treatment Center, Sparta, New Jersey
  - Capital Health Regional Cancer Center, Trenton, New Jersey
  - St. Francis Regional Cancer Center, Trenton, New Jersey
  - Franklin & Edith Scarpa Regional Cancer Center at South Jersey Healthcare, Vineland, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - Lovelace Medical Center - Downtown, Albuquerque, New Mexico
  - Hematology Oncology Associates, PC, Albuquerque, New Mexico
  - New Mexico Cancer Center, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New York Oncology Hematology, PC at Albany Regional Cancer Care, Albany, New York
  - New York Oncology Hematology, PC at Albany Medical Center, Albany, New York
  - Amsterdam Community Cancer Program, Amsterdam, New York
  - Coney Island Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Adirondack Cancer Care - Glens Falls, Glens Falls, New York
  - Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - New York Oncology Hematology, PC - Hudson, Hudson, New York
  - Monter Cancer Center of the North Shore-LIJ Health System, Lake Success, New York
  - New York Oncology Hematology, PC - Latham, Latham, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Northern Westchester Hospital, Mount Kisco, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - Dyson Center for Cancer Care at Vassar Brothers Medical Center, Poughkeepsie, New York
  - Cancer Center of Poughkeepsie, Poughkeepsie, New York
  - Hudson Valley Oncology Associates, Poughkeepsie, New York
  - Saint Francis Hospital Cancer Center, Poughkeepsie, New York
  - Riverview Cancer Care Medical Associates, PC, Rexford, New York
  - Lipson Cancer and Blood Center at Rochester General Hospital, Rochester, New York
  - Interlakes Oncology/Hematology PC, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Nalitt Cancer Institute at Staten Island University Hospital, Staten Island, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Samaritan Hospital at Northeast Health, Troy, New York
  - Dickstein Cancer Treatment Center at White Plains Hospital Center, White Plains, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Hope A Women's Cancer Center, Asheville, North Carolina
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Alamance Cancer Center at Alamance Regional Medical Center, Burlington, North Carolina
  - Waverly Hematology Oncology, Cary, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Batte Cancer Center at Northeast Medical Center, Concord, North Carolina
  - CaroMont Cancer Center at Gaston Memorial Hospital, Gastonia, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Leo W. Jenkins Cancer Center at ECU Medical School, Greenville, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - High Point Regional Hospital, High Point, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Annie Penn Cancer Center, Reidsville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Marion L. Shepard Cancer Center at Beaufort County Hospital, Washington, North Carolina
  - Forsyth Regional Cancer Center at Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - Dakota Cancer Institute at Dakota Clinic - South University, Fargo, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Cleveland Clinic Beachwood Family Health and Surgery Center, Beachwood, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Mercy Cancer Center at Mercy Medical Center, Canton, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Christ Hospital Cancer Center, Cincinnati, Ohio
  - Oncology Hematology Care, Incorporated - Blue Ash, Cincinnati, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center at Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - North Coast Cancer Care - Clyde, Clyde, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Cleveland Clinic Cancer Center, Independence, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - MedCentral - Mansfield Hospital, Mansfield, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Cancer Care Center, Incorporated, Salem, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - United States Air Force Medical Center - Wright-Patterson, Wright-Patterson Air Force Base, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Cleo Craig Cancer Research Clinic, Lawton, Oklahoma
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - St. Charles Medical Center - Bend, Bend, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Three Rivers Community Hospital, Grants Pass, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Dubs Cancer Center at Rogue Valley Medical Center, Medford, Oregon
  - Providence Cancer Center at PMCC, Medford, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center and Children's Hospital, Portland, Oregon
  - Northwest Cancer Specialists at Rose Quarter Cancer Center, Portland, Oregon
  - Kaiser Permanente Health Care - Portland, Portland, Oregon
  - Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Salem Hospital Regional Cancer Care Services, Salem, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Sacred Heart Hospital, Allentown, Pennsylvania
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - St. Luke's Cancer Network at St. Luke's Hospital, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Oncology Hematology Associates of Northern Pennsylvania, PC at Hahne Regional Cancer Center, DuBois, Pennsylvania
  - Dale and Frances Hughes Cancer Center at Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - St. Mary Regional Cancer Center, Langhorne, Pennsylvania
  - Charles A. & Betty Bott Cancer Center at Holy Redeemer Hospital, Meadowbrook, Pennsylvania
  - Riddle Memorial Hospital Cancer Center, Media, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Frankford Hospital Cancer Center - Torresdale Campus, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Cancer Center at Phoenixville Hospital, Phoenixville, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - St. Joseph Medical Center, Reading, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Hematology and Oncology Associates of Northeastern Pennsylvania, Scranton, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Associates in Hematology-Oncology, PC at Crozer Regional Cancer Center, Upland, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Jennersville Regional Hospital, West Grove, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - CCOP - Main Line Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - York Cancer Center at Apple Hill Medical Center, York, Pennsylvania
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Women and Infants Hospital of Rhode Island, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - AnMed Cancer Center, Anderson, South Carolina
  - Roper St. Francis Cancer Center at Roper Hospital, Charleston, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Georgetown Memorial Hospital, Georgetown, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Carolina Blood and Cancer Care Associates, PA, Lancaster, South Carolina
  - Carolina Blood and Cancer Care, Rock Hill, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - U.T. Medical Center Cancer Institute, Knoxville, Tennessee
  - University of Tennessee Cancer Institute - Memphis, Memphis, Tennessee
  - Southwest Regional Cancer Center - Central, Austin, Texas
  - Texas Oncology, PA at Texas Oncology Cancer Center - Central, Austin, Texas
  - Texas Oncology, PA - Austin Northwest, Austin, Texas
  - Texas Oncology, PA - Austin North, Austin, Texas
  - St. Joseph Regional Cancer Center, Bryan, Texas
  - Texas Oncology, PA - Cedar Park, Cedar Park, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Presbyterian Hospital of Dallas, Dallas, Texas
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - UMC Southwest Cancer and Research Center, Lubbock, Texas
  - Texas Oncology, PA - Seton Williamson, Round Rock, Texas
  - Texas Oncology, PA at Texas Cancer Center Round Rock, Round Rock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Texas Oncology, PA - San Marcos, San Marcos, Texas
  - American Fork Hospital, American Fork, Utah
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Lynchburg Hematology-Oncology Clinic, Lynchburg, Virginia
  - Southwest Virginia Regional Cancer Center at Wellmonth Health, Norton, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Carilion Cancer Center of Western Virginia, Roanoke, Virginia
  - Auburn Regional Center for Cancer Care, Auburn, Washington
  - Overlake Cancer Center at Overlake Hospital Medical Center, Bellevue, Washington
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Providence Centralia Hospital, Centralia, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Cascade Cancer Center at Evergreen Hospital Medical Center, Kirkland, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Rockwood Clinic Cancer Treatment Center, Spokane, Washington
  - Cancer Care Northwest - North, Spokane, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - Madigan Army Medical Center - Tacoma, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - St. Mary Regional Cancer Center at St. Mary Medical Center, Walla Walla, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Washington Hematology-Oncology Specialists, Yakima, Washington
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia
  - United Hospital Center, Clarksburg, West Virginia
  - Edwards Comprehensive Cancer Center at Cabell Huntington Hospital, Huntington, West Virginia
  - St. Mary's Regional Cancer Center at St. Mary's Medical Center, Huntington, West Virginia
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - Community Comprehensive Cancer Center at Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - Schiffler Cancer Center at Wheeling Hospital, Wheeling, West Virginia
  - Marshfield Clinic - Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Luther Midlelfort Hospital, Eau Claire, Wisconsin
  - Midelfort Clinic - Luther, Eau Claire, Wisconsin
  - Vince Lombardi Cancer Center at Aurora Lakeland Medical Center - Elkhorn, Elkhorn, Wisconsin
  - Oncology Alliance, SC - Milwaukee - East, Glendale, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Vince Lombardi Cancer Clinic - Green Bay at Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercy Regional Cancer Center, Janesville, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Dean Medical Center - Madison, Madison, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Vince Lombardi Cancer Clinic - Marinette, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Columbia Saint Mary's Hospital - Ozaukee, Mequon, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Columbia-Saint Mary's Cancer Care Center, Milwaukee, Wisconsin
  - Medical Consultants, Limited, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Regional Cancer Center at Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - All Saints Cancer Center at Wheaton Franciscan Healthcare, Racine, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic - Sheboygan, Sheboygan, Wisconsin
  - Saint Michael's Hospital Cancer Center, Stevens Point, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Vince Lombardi Cancer Clinic - Two Rivers, Two Rivers, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
  - Marshfield Clinic - Wausau Center, Wausau, Wisconsin
  - University of Wisconcin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin
  - Aurora Women's Pavilion of West Allis Memorial Hospital, West Allis, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Riverview UW Cancer Center at Riverview Hospital, Wisconsin Rapids, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming
- Canada (18):
  - British Columbia Cancer Agency - Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA - Fraser Valley Cancer Centre, Surrey, British Columbia
  - British Columbia Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia
  - British Columbia Cancer Agency - Vancouver Island Centre, Victoria, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Northeastern Ontario Regional Cancer Centre, Greater Sudbury, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Carlo Fidani Peel Regional Cancer Centre at Credit Valley Hospital, Mississauga, Ontario
  - Cancer Care Program at Thunder Bay Regional Health Sciences, Thunder Bay, Ontario
  - Mount Sinai Hospital - Toronto, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Hopital Notre-Dame du CHUM, Montreal, Quebec
  - CHUM - Hotel Dieu Hospital, Montreal, Quebec
  - CHUM - Hopital Saint-Luc, Montreal, Quebec
  - Royal Victoria Hospital - Montreal, Montreal, Quebec
  - Jewish General Hospital - Montreal, Montreal, Quebec
  - St. Mary's Hospital Center, Montreal, Quebec
  - Hopital du Saint-Sacrement - Quebec, Québec, Quebec
- Ireland (11):
  - Cork University Hospital, Cork
  - South Infirmary Victoria Hospital, Cork
  - Beaumont Hospital, Dublin
  - Adelaide and Meath Hospital, Dublin Incorporating the National Children's Hospital, Dublin
  - St. Vincent's University Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - St. James's Hospital, Dublin
  - University College Hospital, Galway
  - Mid-Western Cancer Centre at Mid-Western Regional Hospital, Limerick
  - Sligo General Hospital, Sligo
  - Waterford Regional Hospital, Waterford

REFERENCES:
- [Background] Mamounas EP, Lembersky B, Jeong JH, Cronin W, Harkins B, Geyer C, Wickerham DL, Paik S, Costantino J, Wolmark N. NSABP B-42: a clinical trial to determine the efficacy of five years of letrozole compared with placebo in patients completing five years of hormonal therapy consisting of an aromatase inhibitor (AI) or tamoxifen followed by an AI in prolonging disease-free survival in postmenopausal women with hormone receptor-positive breast cancer. Clin Breast Cancer. 2006 Dec;7(5):416-21. doi: 10.3816/CBC.2006.n.061. No abstract available. PMID 17239269
- [Derived] Rastogi P, Bandos H, Lucas PC, van 't Veer LJ, Wei JJ, Geyer CE Jr, Fehrenbacher L, Chia SKL, Brufsky AM, Walshe JM, Soori GS, Dakhil SR, Paik S, Swain SM, Menicucci AR, Audeh MW, Wolmark N, Mamounas EP. Utility of the 70-Gene MammaPrint Assay for Prediction of Benefit From Extended Letrozole Therapy in the NRG Oncology/NSABP B-42 Trial. J Clin Oncol. 2024 Oct 20;42(30):3561-3569. doi: 10.1200/JCO.23.01995. Epub 2024 Jul 24. PMID 39047219
- [Derived] Mamounas EP, Bandos H, Lembersky BC, Jeong JH, Geyer CE Jr, Rastogi P, Fehrenbacher L, Graham ML, Chia SK, Brufsky AM, Walshe JM, Soori GS, Dakhil SR, Seay TE, Wade JL 3rd, McCarron EC, Paik S, Swain SM, Wickerham DL, Wolmark N. Use of letrozole after aromatase inhibitor-based therapy in postmenopausal breast cancer (NRG Oncology/NSABP B-42): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2019 Jan;20(1):88-99. doi: 10.1016/S1470-2045(18)30621-1. Epub 2018 Nov 30. PMID 30509771
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 2 Letrozole | Group 1 Placebo
Started | 1983 | 1983
Completed | 1950 | 1953
Not Completed | 33 | 30
Not completed — No follow up data mapped to Other | 17 | 19
Not completed — Patient not at risk for primary endpoint mapped to Other | 7 | 0
Not completed — No clinical assessment | 9 | 11

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo
- Letrozole: Letrozole
- Total: Total of all reporting groups
Arm/Group | Placebo | Letrozole | Total
Number analyzed (Participants) | 1983 | 1983 | 3966
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (8.4) | 63 (8.7) | 63 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1983 | 1983 | 3966
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival
Description: Percentage of patients free from DFS events. DFS events include local, regional, or distant recurrence, second primary cancer or death from any cause prior to recurrence or second primary cancer.
Time Frame: 7 years.
Measure: Number; unit: percentage of patients free of disease
Arm/Group | Group 2 Letrozole | Group 1 Placebo
Number analyzed (Participants) | 1950 | 1953
percentage of patients free of disease | 84.7 | 81.3

2. Secondary Outcome: Overall Survival
Description: Percentage of patients alive
Time Frame: 7 years
Population: Patients with any type of follow up.
Measure: Number; unit: percentage of patients alive
Arm/Group | Group 2 Letrozole | Group 1 Placebo
Number analyzed (Participants) | 1959 | 1964
percentage of patients alive | 91.8 | 92.3

3. Secondary Outcome: Breast Cancer-free Interval
Description: Cumulative incidence of breast-cancer-free interval events. BCFI events include local-regional recurrence, distant recurrence or contralateral breast cancer as a first event.
Time Frame: 7 years
Measure: Number; unit: percentage of patients
Arm/Group | Group 2 Letrozole | Group 1 Placebo
Number analyzed (Participants) | 1950 | 1953
percentage of patients | 6.7 | 10

4. Secondary Outcome: Distant Recurrence
Description: Cumulative incidence of distant recurrences.
Time Frame: 7 years
Measure: Number; unit: percentage of patients
Arm/Group | Group 2 Letrozole | Group 1 Placebo
Number analyzed (Participants) | 1950 | 1953
percentage of patients | 3.9 | 5.8

5. Secondary Outcome: Osteoporotic-related Fractures
Description: Cumulative incidence of osteoporotic-related fractures defined as Colles', hip or spinal fractures
Time Frame: 7 years
Measure: Number; unit: percentage of patients
Arm/Group | Group 2 Letrozole | Group 1 Placebo
Number analyzed (Participants) | 1950 | 1953
percentage of patients | 5.4 | 4.8

6. Secondary Outcome: Arterial Thrombotic Events
Description: Cumulative incidence of arterial thrombotic events, as defined by CTCAE version 4.0 (grade ≥1 stroke or transient ischaemic attack; grade ≥2 acute coronary syndrome or cerebrovascular ischaemia; grade ≥3 myocardial infarction, peripheral ischaemia, or visceral arterial ischaemia; and grade ≥4 selected thromboembolic events [cerebrovascular event, arterial insufficiency]).
Time Frame: 7 years
Measure: Number; unit: percentage of patients
Arm/Group | Group 2 Letrozole | Group 1 Placebo
Number analyzed (Participants) | 1950 | 1953
percentage of patients | 4.0 | 3.4

ADVERSE EVENTS:
Description: Participants at Risk includes any patient who submitted an AE form.
Arm/Group | Placebo | Letrozole
Serious Adverse Events (participants affected / at risk) | 87/1938 | 80/1951
Other Adverse Events (participants affected / at risk) | 336/1938 | 400/1951
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=1938) | Letrozole (N=1951)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alanine aminotransferase increased (ALT/SGPT) (Investigations) | 1 | 2
Amnesia (Nervous system disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 5 | 2
Aortic injury (Injury, poisoning and procedural complications) | 1 | 0
Aspartate aminotransferase increased (AST/SGOT) (Investigations) | 3 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Bladder infection (Infections and infestations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Cardiac arrest (Cardiac disorders) | 3 | 4
Cardiac disorders - Other, specify (Cardiac disorders) | 3 | 2
Cardiac troponin I increased (Investigations) | 2 | 1
Cardiac troponin T increased (Investigations) | 1 | 1
Creatinine increased (Investigations) | 1 | 1
Death NOS (General disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Depression (Psychiatric disorders) | 6 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Encephalopathy (Nervous system disorders) | 2 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 2
Heart failure (Cardiac disorders) | 2 | 5
Hematoma (Vascular disorders) | 1 | 2
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 2
Hypertension (Vascular disorders) | 2 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 4
Hyponatremia (Metabolism and nutrition disorders) | 2 | 1
Hypotension (Vascular disorders) | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 | 1
Intracranial hemorrhage (Nervous system disorders) | 2 | 6
Lipase increased (Investigations) | 0 | 2
Multi-organ failure (General disorders) | 2 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Myocardial infarction (Cardiac disorders) | 9 | 4
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 4
Nervous system disorders - Other, specify (Nervous system disorders) | 3 | 2
Neutrophil count decreased (Investigations) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 1
Personality change (Psychiatric disorders) | 0 | 1
Platelet count decreased (Investigations) | 1 | 1
Psychosis (Psychiatric disorders) | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sepsis (Infections and infestations) | 2 | 4
Serum amylase increased (Investigations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Stroke (Nervous system disorders) | 2 | 2
Suicidal ideation (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 1
Thromboembolic event (Vascular disorders) | 8 | 1
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 4
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Leukemia secondary to oncology chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
White blood cell decreased (Investigations) | 0 | 1
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Mediastinal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Right ventricular dysfunction (Cardiac disorders) | 1 | 0
Lung infection (Infections and infestations) | 6 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Aortic valve disease (Cardiac disorders) | 5 | 3
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Soft tissue necrosis lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 2
Left ventricular systolic dysfunction (Cardiac disorders) | 2 | 6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=1938) | Letrozole (N=1951)
Arthralgia (Musculoskeletal and connective tissue disorders) | 302 | 347
Myalgia (Musculoskeletal and connective tissue disorders) | 118 | 149

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less